CLINICAL TRIAL: NCT06524687
Title: A Phase 1b, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Imvotamab in Adult Participants With Active, Refractory Moderate-Severe Idiopathic Inflammatory Myopathies
Brief Title: A Study of Imvotamab in Active, Refractory Idiopathic Inflammatory Myopathies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Program Discontinuation
Sponsor: IGM Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGM-2323-103
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Inflammatory Myopathies; Inflammatory Myopathies
Keywords: Myopathies; Moderate-Severe Myopathy; Myositis
MeSH Terms: conditions — Myositis; Muscular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imvotamab (Dose Escalation) (Experimental): Imvotamab administered intravenously
  Interventions: Drug: Imvotamab

INTERVENTIONS:
Drug: Imvotamab — Administered intravenously

SUMMARY:
The purpose of this study is to determine the safety and tolerability of imvotamab in patients with Moderate-Severe Idiopathic Inflammatory Myopathies who have failed prior therapies.

Participants will be given imvotamab through a vein (i.e., intravenously).

DETAILED DESCRIPTION:
This is a Phase 1b, open-label study to determine the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of imvotamab in adult participants with active, refractory, moderate-severe Idiopathic Inflammatory Myopathies. Approximately 5-10 participants will be assigned.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years at the time of signing ICF
* Diagnosis of probable or definite IIM according to the 2017 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for IIM with subgroup classification of either DM, polymyositis (PM), anti-synthetase syndrome, or immune-mediated necrotizing myositis (IMNM).
* Active IIM despite treatment with corticosteroids and at least 1 immunosuppressive or immunomodulatory standard-of-care agent determined at the discretion of the investigator after at least 3 months of treatment.
* If using oral corticosteroids (OCS), must be on a stable dose equivalent to ≤ 30 mg/day of prednisone for at least 4 weeks prior to first study treatment

Key Exclusion Criteria:

* Pregnant or breastfeeding or intending to become pregnant during the study or within 3 months after the final dose of imvotamab.
* Receipt of an investigational therapy less than 12 weeks or 5 drug-elimination half-lives (whichever is longer) prior to first administration of study treatment and during the study.
* Has inclusion body myositis or myositis-associated with other connective tissue disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of imvotamab | Time Frame: Up to Week 50
  Incidence of adverse events (AEs), serious adverse events (SAEs), including serious

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kunder, Study Director — IGM Biosciences
Locations (1):
- Standford University, Palo Alto, California, United States